CLINICAL TRIAL: NCT04840069
Title: A Phase II Randomized Clinical Trial of Radiotherapy Planning Using Conventional Imaging +/- Fluciclovine PET in Patients With Newly Diagnosed Glioblastoma
Brief Title: Radiotherapy Planning Using Fluciclovine PET in Patients With Newly Diagnosed Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Foundation (Other); Arizona Biomedical Research Commission (ABRC) (Other); Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090-20-16
Record Dates: First submitted 2021-03-16; First posted 2021-04-09 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MRI-guided radiotherapy (No Intervention): Patients will undergo standard of care MRI-guided radiotherapy.
- MRI + Fluciclovine PET-guided radiotherapy (Experimental): Patients will undergo MRI + Fluciclovine PET-guided radiotherapy
  Interventions: Drug: Fluciclovine PET guided Radiotherapy

INTERVENTIONS:
Drug: Fluciclovine PET guided Radiotherapy — PET+MRI Based There is no GTV_5400. The GTV_6000 will be defined as the surgical cavity inclusive of any remaining tumor enhancement and the hypermetabolic volume. CTV_5400 will include the GTV_6000 plus a margin of 1.0 cm which may be reduced around natural barriers to tumor growth such as the skull, ventricles, falx, etc. CTV_5400 must also include the entirety of the GTV_6000. There is no CTV_6000. PTV_5400 is the CTV_5400 plus a geometric 3 mm expansion in all dimensions; PTV_6000 is GTV_6000 plus a geometric 3 mm expansion in all dimensions. PTV may extend beyond bony margins and the skin surface. The PTV_5400 must contain the PTV_6000. In the setting of multi-focal disease, the primary target volumes will be defined as above, but for satellite lesions, the GTV_6000 will be defined as any tumor enhancement and hypermetabolic volume. There will be no CTV_6000. PTV_6000 will be defined as GTV_6000 plus a geometric 3 mm expansion in all dimensions.
  Arms: MRI + Fluciclovine PET-guided radiotherapy

SUMMARY:
The purpose of the this study is to see if the use of a PET scan with 18F-fluciclovine (PET or Fluciclovine PET) in addition to the normal radiation planning imaging procedures (MRI and CT scan) will help determine the areas where the radiation therapy is to be delivered. It is also a goal of the study to determine if subjects live longer when treatment plans for radiation therapy are designed using a Fluciclovine PET scan, as well as MRI and CT scans. We will also collect information on if and where the tumor returns. Information on the side effects from the two different treatment planning imaging methods will also be collected. 18F-Fluciclovine is an FDA-approved radioactive diagnostic agent that is injected into the patient and then taken up by cancer cells, which can then be visualized with a PET/CT scan. 18F-Fluciclovine is FDA approved for the detection of recurrent prostate cancer, but is still investigational for the purposes of this study.

DETAILED DESCRIPTION:
The goal of this study is to see if the use of PET in planning radiotherapy can reduce these local failures.

Glioblastoma (GBM) is the most common primary malignant brain tumor. Newly diagnosed glioblastoma management includes maximum safe resection followed by radiotherapy with concurrent temozolomide, followed by maintenance temozolomide for 6 - 12 cycles. This postoperative chemoradiotherapy approach has resulted in a significant increase in median PFS (5.0 vs. 6.9 months) and OS (12.1 vs. 14.6 months) compared to radiotherapy alone (Stupp 2005). However, despite such multi-modality therapy, the median survival for GBM remains poor at approximately 15-16 months in contemporary series (Grossman, Ye et al. 2010, Gilbert, Wang et al. 2013 vs 2010).

Recently, a randomized trial of tumor-treating fields (TTF or Optune) plus temozolomide demonstrated the benefit of this treatment in newly diagnosed glioblastoma that led to FDA approval of the device (Stupp 2015, Stupp 2017). However despite these advances, most patients still have a poor prognosis with median survival of 16-21 months. Although adjuvant chemoradiotherapy has been shown to increase survival, a predominant pattern of failure remains local (Chan, Lee et al. 2002, Milano, Okunieff et al. 2010). Therefore, better therapeutic options are needed for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary, newly diagnosed supratentorial, WHO grade IV glioma
* Greater than 18 years of age
* Karnofsky performance score greater than 70%
* Recovered from surgery and on a stable or tapering dose of corticosteroids
* Plan to undergo standard therapy with XRT 60Gy/30fx with TMZ followed by 6-12 cycles of maintenance TMZ within 6 weeks of surgery
* If woman of child bearing potential, negative serum pregnancy test. Patients must agree to take adequate pregnancy preventions for the length of the study.
* Life expectancy of at least 3 months
* Written study specific consent

Exclusion Criteria:

* Previous treatment of glioma of any grade with bevacizumab or other molecular targeted therapies less than 6 months before MRI (and PET) used for radiotherapy planning
* Recurrent of multifocal malignant glioma
* Any sites of distant disease (for example drop metastases or leptomeningeal spread)
* Prior use of Gliadel wafers or any other intratumal or intracavity treatment
* Prior radiotherapy to the cranium, head and neck or other sites resulting in overlapping fields
* Molecular targeted therapies planned during radiotherapy
* Simultaneous participation in other interventional trials which could interfere with this trial or participation in a clinical trial within the last thirty days before patient's enrollment in current study.
* Inability to undergo an MRI or PET (Claustrophobia, non-MRI compatible pacemaker, known allergy to MRI contrast agent or fluciclovine tracer)
* Any pregnant or lactating patient
* Any prior malignancy within 3 years excluding carcinoma in-situ or early staged,localized basal or squamous cell skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Patterns of Failure | 36 months
  To assess whether incorporating fluciclovine PET into radiotherapy planning significantly changes the in-field and out-of-field radiographic progression rates, by comparison to traditional MRI-based radiotherapy
Defining Tumor Volume | 36 months
  2. To determine the effect fluciclovine PET has on definition of the tumor volume, as compared to traditional MRI-based radiotherapy.

SECONDARY OUTCOMES:
Survival using MRI radiotherapy | 36 months
  To quantify overall and progression free survival utilizing MRI cohort.
Overall survival utilizing MRI+PET radiotherapy | 36 months
  To quantify overall survival utilizing MRI+PET-based radiotherapy
Progression free survival utilizing MRI+PET-based radiotherapy | 36 months
  To quantify progression free survival utilizing MRI+PET-based

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States